CLINICAL TRIAL: NCT02903303
Title: Pilot Study : Hypnosis as a Potentiation Technique for the Interventional Treatment of Chronic Lumbar Pain
Brief Title: Hypnosis as a Potentiation Technique for the Interventional Treatment of Chronic Lumbar Pain
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: end of recruitment period
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, Marc R Suter, PD Doctor, Centre Hospitalier Universitaire Vaudois
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-00236
Record Dates: First submitted 2016-05-27; First posted 2016-09-16 (Estimated); Last update posted 2021-08-23 (Actual); Status verified 2021-08

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain | interventions — Hypnosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Other): There will be only one arm for this pilot study. All participants will follow 4 hypnosis sessions, and then the facet block.
  Interventions: Other: Hypnosis

INTERVENTIONS:
Other: Hypnosis — It will consist in 4 hypnosis sessions within 2 weeks mainly for analgesic purpose. The main themes are :
  * 1st session : contact with the therapist, body scan, basic suggestions
  * 2nd session : hypnosis induction followed by suggestions tu build a safe place
  * 3rd session : it is the first complete hypnosis session (induction and specific suggestions against pain)
  * 4th session : very similar to the previous session for the content, focused on auto-hypnosis learning.

SUMMARY:
This pilot study consists in testing the efficacy of hypnosis as an adjuvant treatment for patients suffering from chronic lumbar pain and for whom a facet block is indicated by a doctor in the Centre d'antalgie of CHUV (Centre Hospitalier Universitaire Vaudois), where this study will take place. 5 to 8 patients will be included in this study. The goals of this study are :

* Assess the feasibility of such a protocol with more patients
* Measure the number of patients necessary to obtain a significant result
* Search for possible side effects of the combination of both treatments

Every patient in this pilot study will undergo 4 hypnosis sessions within 2 weeks before the facet block. These sessions will be done with an hypnotherapist formed for this kind of treatment.

Three times during this study, each patient will have a discussion with the co-investigator :¨

* 1st discussion : just before the first hypnosis session
* 2nd discussion : after the 4 hypnosis sessions and just before the facet block, approximately 3 to 4 weeks after the 1st discussion
* 3rd discussion : 2 to 4 weeks after the facet block

They will allow to obtain several data :

* Pain assessment : intensity, localization, variability, characteristics, effects on daily life activities
* Anxiety and depression assessment
* Expectations assessment : about both treatments and their combination
* Efficacy assessment : about both treatments for the patient
* Questions about the perceptions of the treatments (prejudice, ...) et possible side effects.

These data will then be analysed (quantitative and qualitative analysis, depending on the question type) to fulfill the objectives of the study.

will include 5 to 8 people suffering from chronic lumbar pain. The procedure consists in two steps :

1. 4 hypnosis sessions as an adjuvant treatment for number 2
2. a facet block, which is the standard procedure in the Centre d'antalgie in CHUV.

There will be no control group, so every patient will participate to the hypnosis sessions and undergo the facet block. All the procedure of the facet block (including contraindications and side effects) are not considered to be part of this study because all patients in this study would have had a facet block if they would not participate in it.

The only data that will be collected are questionnaires about several items (pain, anxiety, depression, ...). These questionnaires are filled with the patient at the beginning of the study (day 0), before the facet block (between day 14 and day 21) and 2-4 weeks after it (between day 28 and day 49). There are quantitative and qualitative questions.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent and signature of the declaration of consent ;
* Patient suffering from chronic lumbar pain (> 3 months)
* Indication for a facet block ;
* Good ability to speak and understand French.

Exclusion Criteria:

* Previous facet block for the same indication ;
* Unability to understand or speak French ;
* Unability to understand the written or oral instructions necessary to the protocol application ;
* Acute or severe psychiatric decompensation and/or acute psychosocial distress ;
* Complex psychosocial situation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2016-09-01 (Actual); Study Completion 2016-09-01 (Actual)

PRIMARY OUTCOMES:
Daily pain history | 1st encounter with the co-investigator (day 0)
  During the first encounter (day 0), we will ask the patient since when he/she suffers from daily pain:
  * Daily pain in general since : < 3 months ; 3-6 months ; 6-12 months ; 1-3 years ; 3-5 years ; 5-10 years ; 10-20 years ; > 20 years
  * Daily lumbar pain since : < 6 months ; 6-12 months ; 1-3 years ; > 3 years
Change in pain localization | 1st, 2nd and 3rd encounters with the co-investigator (day 0, day 14-21, day 28-49)
  For this outcome, the patient is asked to say where is the daily pain and to precise if the pain concerns both sides. If there is more than one localization, the patient is asked to say which pain is the worst for him/her.
Change in neuropathic characteristics of the lumbar pain | 1st, 2nd and 3rd encounters with the co-investigator (day 0, day 14-21, day 28-49)
  Neuropathic characteristics (yes/no) :
  * burning
  * painful cold
  * electricity sensation
  * swarming
  * tingle
  * itching
  * numbness
Change in lumbar pain intensity | 1st, 2nd and 3rd encounters with the co-investigator (day 0, day 14-21, day 28-49)
  Intensity on a scale from 0 (no pain) to 10 (worst pain imaginable) :
  * Worst pain during the previous week
  * Lowest pain during the previous week
  * Average pain during the previous week
Change in lumbar pain interferences | 1st, 2nd and 3rd encounters with the co-investigator (day 0, day 14-21, day 28-49)
  For this outcome, we will ask the patient to tell us how much between 0 (no influence at all) and 10 (complete discomfort) the lumbar pain has on :
  A) General activity B) Mood C) Ability to walk D) Usual work E) Relationship with others F) Sleep G) Taste of living
Change in Anxiety and Depression assessment | 1st and 3rd encounters with the co-investigator (day 0, day 28-49)
  In this pilot study, we will use the HADS scale (Hospital Anxiety and Depression Scale) to assess the level of anxiety and depression at the beginning of the study (day 0) and at the end of it (day 28-49). The items are the following (on a scale from 0 to 3, depending on the agreement to the sentence) :
  1. I feel tense and angry
  2. I am afraid, just like if something horrible was going to happen to me
  3. I'm worried
  4. I can sit quietly doing nothing and feel relaxed
  5. I experience feelings of fear and feel my stomach tensed
  6. I have ants in my pants and can't stay in place
  7. I experience sudden feelings of panic
  8. I feel the same pleasure to the same things as before
  9. I easily laugh and see things in a good way
  10. I am in a good mood
  11. I feel like I work slowly
  12. I don't take care about my appearance anymore
  13. I'm looking forward to doing some things
  14. I can enjoy a good book or a good TV/radio show
Presumed efficacy and expectations about treatments of lumbar pain | 1st encounter (day 0)
  On a scale from 0 (no efficacy at all) to 10 (completely relieves the pain), the patient assesses the presumed efficacy in general of : (only for the 1st encounter)
  1. Hypnosis alone
  2. Facet block alone
  3. Combination of both
  On a scale from 0 to 10, the patient assesses the expectations towards 1), 2) and 3).
Efficacy about treatments of lumbar pain | 3rd encounter (day 28-49)
  On a scale from 0 (no efficacy at all) to 10 (completely relieves the pain), the patient assesses the efficacy of :
  1. Hypnosis alone
  2. Facet block alone
  3. Combination of both
Functionality enhancement expectations thanks to hypnosis | 1st encounter (day 0)
  On a scale from 1 (minimal impact) to 5 (maximal enhancement), the patient assesses how much he/she thinks hypnosis will enhance the ability to :
  1. do sports
  2. practice the professional activity
  3. do your daily activities
  4. enhance your mood
  5. other (free space for the patient to write)
Functionality enhancement thanks to hypnosis | 3rd encounter (day 28-40)
  On a scale from 1 (minimal impact) to 5 (maximal enhancement), the patient assesses how much hypnosis has enhanced his/her ability to :
  1. do sports
  2. practice the professional activity
  3. do your daily activities
  4. enhance your mood
  5. other (same item as in outcome 9)
Questions with a qualitative analysis (part 1) | 1st encounter (day 0)
  During this encounter, we will ask questions to the patient and write down the main subjects mentioned, so that a theme-based analysis can be done with these. The questions are the following :
  * How do you think hypnosis work ?
  * What do you think will happen during hypnosis ?
  * Does it make you experience any emotions ?
  * What do you think of hypnosis as a therapeutical approach ?
  * How do you think facet block works ?
  * What do you think will happen during this intervention ?
  * What do you think of facet block as a therapeutical approach ?
  * What is your position about pain-relief drugs ?
  * Do you use other approaches against pain ? If yes, which one and what does and doesn't work with you ?
  * Do you have further comments about both treatments ?
Questions with a qualitative analysis (part 2) | 3rd encounter (day 28-49)
  During this encounter, we will ask questions to the patient and write down the main subjects mentioned, so that a theme-based analysis can be done with these. The questions are the following :
  * How do you feel now about hypnosis as a treatment against pain ?
  * Did your mind change about hypnosis ? If yes, how and in what ?
  * Now, do you consider using hypnosis and/or self-hypnosis as a new way to deal with your lumbar pain ?
  * Do you have further comments about the study or the procedure ?

SECONDARY OUTCOMES:
Security assessment | 2nd and 3rd encounters (day 14-21, day 24-49)
  Immediately after the beginning of the study, every patient will be told to report every adverse effect or discomfort during or after an hypnosis session. During the hypnosis session, the therapist will be vigilant about possible negative effects and will help the patient go through it. He will also make a report about it.
  Every adverse effect will be discussed in detail with the patient during the 2nd or the 3rd discussion with the co-investigator.

CONTACTS AND LOCATIONS:
Overall Officials: Marc Suter, Doctor, PD, Principal Investigator — Centre Hospitalier Universitaire Vaudois
Locations (1):
- Centre d'antalgie, Centre Hospitalier Universitaire Vaudois, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: No
Participant data will remain accessible only for the people working in this study. However, the results will be shown in the context of a master degree in medicine of Mr Florent Schroeter.